CLINICAL TRIAL: NCT01400724
Title: Effects of Inofolic NRT on Post-menopausal Women Affected by the Metabolic Syndrome
Brief Title: Inofolic NRT and the Metabolic Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Messina (Other)
Responsible Party: Principal Investigator, Rosario D'anna, associate professor, University of Messina
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: INOFOLIC-NRT; NRT-LO.LI (Other Grant/Funding Number: LO.LI Pharma)
Record Dates: First submitted 2011-07-14; First posted 2011-07-22 (Estimated); Last update posted 2013-07-16 (Estimated); Status verified 2013-07

CONDITIONS: Metabolic Syndrome; Postmenopausal Disorder
Keywords: menopause; metabolic syndrome; myo-inositol; insulin resistance; cocoa polyphenols; isoflavones
MeSH Terms: conditions — Metabolic Syndrome; Insulin Resistance

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (1):
- Inofolic NRT (Experimental)
  Interventions: Dietary Supplement: Inofolic NRT

INTERVENTIONS:
Dietary Supplement: Inofolic NRT — Dietary supplement: myo-inositol 2000 mg plus cocoa polyphenols 30 mg and plus isoflavones 80 mg

SUMMARY:
A prospective, randomized, controlled, open-label study will be carried out on 80 post-menopausal women affected by the metabolic syndrome (criteria are described in NIH ATP III). After a written informed consent, women will be randomly treated for 6 months with hypocaloric diet (control group) or with diet and a supplementation of myo-inositol 2000 mg plus cocoa polyphenols 30 mg and plus isoflavones 80 mg. will be given randomly Eighty post-menopausal women, affected by metabolic syndrome will be randomized into two groups: 40 treated with myo-inositol 2 g twice per day and forty treated with placebo for six months. The investigators hypothesize that the administration of myo-inositol would improve the insulin-receptor activity in these women, reducing insulin resistance.

DETAILED DESCRIPTION:
Inclusion Criteria: post-menopausal women (12 months after last menstruation) affected by metabolic syndrome according to ATP III, 2001.

At least 3 of following 5 criteria must be present:

1. waist circumference > 88 cm
2. Triglycerides > 150 mg/dl
3. HDL-cholesterol < 50 mg/dl
4. Fast glycemia > 110 mg/dl
5. Systolic blood pressure > 135 mmHg. diastolic > 85 mmHg -

Exclusion Criteria:1) post-menopausal women with less than 12 months from the last menstruation 2) less than 3 criteria according with ATP III 3) TSH > 3.5 4) in treatment with drugs lowering glycemia or cholesterol 5) allergy to cocoa

ELIGIBILITY:
Inclusion Criteria: post-menopausal women (12 months after last menstruation) affected by metabolic syndrome according to ATP III, 2001.

At least 3 of following 5 criteria must be present:

1. waist circumference > 88 cm
2. Triglycerides > 150 mg/dl
3. HDL-cholesterol < 50 mg/dl
4. Fast glycemia > 110 mg/dl
5. Systolic blood pressure > 135 mmHg. diastolic > 85 mmHg -

Exclusion Criteria:

1. post-menopausal women with less than 12 months from the last menstruation
2. less than 3 criteria according with ATP III
3. TSH > 3.5
4. in treatment with drugs lowering glycemia or cholesterol
5. allergy to cocoa

Ages: 50 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2011-06; Primary Completion 2012-07 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
percentage reduction of women with metabolic syndrome | at baseline and after 6 months.
  evaluation of metabolic syndrome criteria according with ATP III 2001

SECONDARY OUTCOMES:
reduction of insulin resistance | at baseline and after 6 months
  evaluation of HOMA-IR
Improvement of lipid profile | at baseline and after 6 months
  reduction of serum triglycerides and increase of HDL-cholesterol
variation in serum concentration of adiponectin, visfatin and resistin | at baseline and after 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Rosario D'Anna, professor, Principal Investigator — University of Messina
Locations (1):
- University Hospital, Messina, Italy

REFERENCES:
- [Derived] D'Anna R, Santamaria A, Cannata ML, Interdonato ML, Giorgianni GM, Granese R, Corrado F, Bitto A. Effects of a new flavonoid and Myo-inositol supplement on some biomarkers of cardiovascular risk in postmenopausal women: a randomized trial. Int J Endocrinol. 2014;2014:653561. doi: 10.1155/2014/653561. Epub 2014 Aug 31. PMID 25254044